CLINICAL TRIAL: NCT02525835
Title: Tissue Sodium in Autoimmune Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine and Pharmacology, Assc. Director Division of Clinical Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 150713
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dietary Sodium (Experimental): Participants will be randomized to a low sodium diet (50 mmol/24 hours) for 28 days (range allowed 25-31 days) or a high sodium diet (250 mmol/24 hours) for 28 days (range allowed 25-31 days) with a 4 week washout period between (range 2-3 weeks).
  Interventions: Dietary Supplement: Low Dietary Sodium
- High Dietary Sodium (Experimental): Participants will be randomized to a low sodium diet (50 mmol/24 hours) for 28 days (range allowed 25-31 days) or a high sodium diet (250 mmol/24 hours) for 28 days (range allowed 25-31 days) with a 4 week washout period between (range 2-3 weeks).
  Interventions: Dietary Supplement: High Dietary Sodium

INTERVENTIONS:
Dietary Supplement: Low Dietary Sodium — Participants will be randomized to a low sodium diet (50 mmol/24 hours) for 28 days (range allowed 25-31 days) with a 4 week washout period between (range 2-3 weeks).
  Arms: Low Dietary Sodium
Dietary Supplement: High Dietary Sodium — Participants will be randomized to a high sodium diet (250 mmol/24 hours) for 28 days (range allowed 25-31 days) with a 4 week washout period between (range 2-3 weeks).
  Arms: High Dietary Sodium

SUMMARY:
This pilot study will test the hypothesis that a low sodium diet will decrease sodium (23Na) magnetic resonance imaging-determined skin sodium concentrations in patients with systemic lupus erythematosus (SLE) and improve blood pressure and inflammation

DETAILED DESCRIPTION:
This pilot study will test the hypothesis that a low sodium diet will decrease 23Na magnetic resonance imaging-determined skin sodium concentrations in patients with SLE and improve blood pressure and inflammation. Investigators plan to enroll 21 participants who will be randomized to low salt or high salt diet. Participants will eat the first diet for 28 days, and after a 2 week washout, Participants will eat the second diet (whichever the participant was not randomized to for the first phase). Participant will know what diet participant is on, study coordinator who does the assessment will be blinded to diet.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients 18 and over
* meets 2012 International criteria for the diagnosis of SLE
* have stable disease activity as evidenced by no significant change in immunomodulating therapy in last month
* provide written informed consent

Exclusion Criteria:

* Pregnancy
* Receiving dialysis
* Organ or bone marrow transplant
* Uncontrolled hypertension, BP> 160/100 mm Hg at screening
* Severe edema as judged by investigator
* Diabetes mellitus requiring drug therapy
* Major surgery within the previous 3 months
* Severe co-morbid conditions such as active cancer likely to compromise study participation
* unwillingness or other inability to cooperate
* Conditions that alter sodium homeostasis substantially including heart failure, clinically evident liver disease, clinically evident renal dysfunction (creatinine clearance < 50 nl/min or > 2+ proteinuria, or being treated for lupus nephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
sodium concentration in skin | 3 months
  sodium concentration in skin after 1 month low salt diet will be compared to sodium concentration in skin after 1 month high sodium diet, with 2 week wash out between

SECONDARY OUTCOMES:
SLEDAI | 3 months
  SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index, a list of 24 items that covers clinical findings and laboratory tests that combined indicate how active a participant's disease is. SLEDAI after 1 month low salt diet will be compared to SLEDAI after 1 month high sodium diet, with 2 week wash out between
blood pressure | 3 months
  Blood pressure after 1 month low salt diet will be compared to blood pressure after 1 month high sodium diet, with 2 week wash out between

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Stein, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States